CLINICAL TRIAL: NCT01103609
Title: An Open-Label, Randomised, Placebo-Controlled, Two-Way Crossover, Phase I Single Centre Study in Type 2 Diabetes Mellitus Patients Treated With Metformin to Evaluate the Pharmacokinetics and Pharmacodynamics of Warfarin During Co-administration With AZD1656
Brief Title: Investigate the Effect of AZD1656 on the Pharmacokinetics and Pharmacodynamics of Warfarin in Type 2 Diabetes Mellitus (T2DM) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1020C00027
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; Type 2; Warfarin; drug-drug interaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Warfarin; AZD1656

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): twice daily on Day 1 to Day 10, with Warfarin on Day 4
  Interventions: Drug: Warfarin; Drug: AZD1656
- 2 (Placebo Comparator): twice daily on Day 1 to Day 10, with Warfarin on Day 4
  Interventions: Drug: Warfarin; Drug: Placebo

INTERVENTIONS:
Drug: Warfarin — Oral tablet od on Day 4
Drug: Placebo — Oral tablet bd, stepwise increased
  Arms: 2
Drug: AZD1656 — Oral tablet bd, stepwise increased
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether AZD1656 will affect the Pharmacokinetics and Pharmacodynamics of Warfarin in T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of T2DM treated with at least 1000 mg metformin as a single treatment or in combination with one other oral anti-diabetics for at least 2 months prior to screening. Doses of anti-diabetic treatment stable for at least 1 month
* Fasting plasma glucose (FPG) at screening in the range of 6.0 to 15.0 mmol/L (108 to 270 mg/dL) and FPG in the range of 7.5 to 13.0 mmol/L (135 to 234 mg/dL) on Day 1
* Haemoglobin (Hb) A1c >6.5% at screening

Exclusion Criteria:

* Use of drugs with anticoagulant effects 3 weeks prior to first warfarin dosing
* Use of amiodarone within 3 months prior to screening and the use of potent CYP450 inhibitors
* Previous treatment with warfarin on clinical indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of warfarin after a single dose when administered alone and in combination with AZD1656 at steady state by assessment of AUC and Cmax of both enantiomers of warfarin (S- and R-warfarin). | Serial PK blood samples will be taken on days 4-10 during the treatment periods

SECONDARY OUTCOMES:
To evaluate the anticoagulant activity of warfarin upon co-administration with AZD1656 by assessment of prothrombin time (PT) and international normalised ratio (INR). | Serial blood samples for warfarin PD measurements will be taken on days 4-10 during the treatment periods
To evaluate the safety of AZD1656 in combination with warfarin by assessment of electrocardiogram, weight, pulse, blood pressure, laboratory variables (including 7-point glucose), physical examination and adverse events | Safety assessments will be monitored throughout the study, from screening visit until follow up visit.
To describe the pharmacokinetics of AZD1656 and its metabolite during concomitant warfarin administration by assessment of AUC0-24, Cmax, Ctrough, tmax, t1/2 and CL/F (AZD1656 only). | Serial PK blood samples will be taken on days 4-10 during the treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Stanko Skrtic, Study Director — AstraZeneca; James Ritter, Prof, Principal Investigator — Quintiles Drug Research Unit; Mirjana Kujacic, Study Chair — AstraZeneca
Locations (1):
- Research Site, London, United Kingdom